CLINICAL TRIAL: NCT01967784
Title: Immunogenicity and Safety of a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route in Children and Adolescents in Taiwan
Brief Title: Study of a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route in Children and Adolescents in Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GQM09; U1111-1127-7693 (Other: WHO)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Influenza
Keywords: Influenza; Quadrivalent Inactivated Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Participants age 9 to 17 years will receive a dose of Quadrivalent Influenza Vaccine
  Interventions: Biological: Quadrivalent Influenza Vaccine (split virion, inactivated)

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine (split virion, inactivated) — 0.5 mL, Intramuscular

SUMMARY:
The aim of the study is to describe the immunogenicity and safety of the new formulation of Quadrivalent Influenza Vaccine (QIV) for the 2013-2014 season in the Northern Hemisphere (NH) in subjects aged 9 to 17 years in Taiwan

Primary Objective:

* To describe the immunogenicity of the QIV (split-virion, inactivated) NH seasonal formulation

Secondary Objective:

* To describe the safety of the QIV (split-virion, inactivated) NH seasonal formulation

DETAILED DESCRIPTION:
Study participants will be vaccinated with one dose of the QIV (split-virion, inactivated) NH 2013-2014 formulation by the intramuscular route or deep subcutaneous. Immunogenicity will be assessed at baseline (Day 0) and 21 days after injection; they will also be followed-up for safety for 21 days after injection.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 to 17 years on the day of inclusion
* Assent form (AF) and/or informed consent form (ICF) have been signed and dated by the subject according to each site requirements, and ICF has been signed and dated by the parent(s) or another legally acceptable representative(s) and by an independent witness if applicable
* Subject and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Subject is pregnant (or positive urine pregnancy test), or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination)
* Participation at the time of study enrollment or in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 3 weeks following trial vaccination
* Vaccination against influenza in the previous 12 months if administered in the context of a clinical trial or in the previous 6 months if administered in the context of a flu vaccination campaign
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported history of seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C, after questioning
* Known systemic hypersensitivity to eggs, chicken proteins, neomycin, formaldehyde and octoxynol-9, or to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the study or to a vaccine containing any of the same substances
* Known or suspected thrombocytopenia, contraindicating intramuscular vaccination based on investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination upon investigator's judgment
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥38.0°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as a family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (2):
- Taiwan (2):
  - Taipei
  - Taoyuan District

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 18 October 2013 to 19 November 2013 at 2 clinical sites in Taiwan.
Pre-assignment Details: A total of 100 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and vaccinated in the study.
Groups:
- Quadrivalent Influenza Vaccine: Participants aged 9 to 17 years of age who received one dose of the quadrivalent influenza vaccine (QIV) (split-virion, inactivated) Northern Hemisphere (NH) 2013-2014 formulation.
Period: Overall Study
Arm/Group | Quadrivalent Influenza Vaccine
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 13.4 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 54
Region of Enrollment [Number; unit: Participants]
  Taiwan | 100

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers of Influenza Antibodies Before and Following Vaccination With a Quadrivalent Influenza Vaccine
Description: Immunogenicity of the Quadrivalent Influenza Vaccine virus was evaluated using the hemagglutination inhibition (HAI) technique.
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Geometric mean titers were analyzed in the Immunogenicity Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 100
Titers (1/dilution)
  A/California/07/2009 (H1N1); Pre-dose | 257 [204 to 324]
  A/California/07/2009 (H1N1); Post-dose | 589 [498 to 697]
  A/Texas/50/2012 (H3N2); Pre-dose | 382 [301 to 484]
  A/Texas/50/2012 (H3N2); Post-dose | 782 [649 to 944]
  B/Massachusetts/2/2012; Pre-dose | 497 [366 to 674]
  B/Massachusetts/2/2012; Post-dose | 1654 [1352 to 2024]
  B/Brisbane/60/2008; Pre-dose | 186 [139 to 250]
  B/Brisbane/60/2008; Post-dose | 856 [702 to 1045]

2. Primary Outcome: Percentage of Participants With Seroprotection Before and Following Vaccination With a Quadrivalent Influenza Vaccine
Description: Immunogenicity of the Quadrivalent Influenza vaccine virus was evaluated using the hemagglutination inhibition (HAI) technique. Seroprotection was defined as titers ≥ 40 (1/dil) on Day 0 (pre-vaccination) and on Day 21 post-vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Seroprotection was analyzed in the Immunogenicity Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 100
Percentage of participants
  A/California/07/2009 (H1N1); Pre-dose | 95.0
  A/California/07/2009 (H1N1); Post-dose | 100.0
  A/Texas/50/2012 (H3N2); Pre-dose | 97.0
  A/Texas/50/2012 (H3N2); Post-dose | 99.0
  B/Massachusetts/2/2012; Pre-dose | 94.0
  B/Massachusetts/2/2012; Post-dose | 100.0
  B/Brisbane/60/2008; Pre-dose | 85.0
  B/Brisbane/60/2008; Post-dose | 100.0

3. Primary Outcome: Percentage of Participants With Seroconversion or Significant Increase in Influenza Antibody Titers Following Vaccination With a Quadrivalent Influenza Vaccine
Description: Immunogenicity of the Quadrivalent Influenza vaccine virus was evaluated using the hemagglutination inhibition (HAI) technique. Seroconversion was defined as participants with a pre-vaccination titer <10 (1/dil) to a post-vaccination titer ≥40 (1/dil) or significant increase was defined as participants with a pre-vaccination titer ≥10 (1/dil) and ≥4-fold increase of the titer.
Time Frame: Day 21 post-vaccination
Population: Seroconversion or significant increase in influenza antibody titers was analyzed in the Immunogenicity Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 100
Percentage of participants
  A/California/07/2009 (H1N1) | 24.0
  A/Texas/50/2012 (H3N2) | 20.0
  B/Massachusetts/2/2012 | 39.0
  B/Brisbane/60/2008 | 48.0

4. Primary Outcome: Geometric Mean Titers Ratios of Influenza Antibodies Following Vaccination With a Quadrivalent Influenza Vaccine
Description: as for outcome 1
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Geometric mean titers ratios were analyzed in the Immunogenicity Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers ratio
Arm/Group | Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 100
Titers ratio
  A/California/07/2009 (H1N1) | 2.29 [1.93 to 2.71]
  A/Texas/50/2012 (H3N2) | 2.05 [1.76 to 2.39]
  B/Massachusetts/2/2012 | 3.33 [2.57 to 4.31]
  B/Brisbane/60/2008 | 4.59 [3.63 to 5.81]

5. Primary Outcome: Percentage of Participants Reporting Solicited Injection Site or Systemic Reactions Following Vaccination With a Quadrivalent Influenza Vaccine
Description: Solicited Injection site: Pain, Erythema, Swelling, Induration, and Ecchymosis. Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Shivering. Injection site Grade 3 (9 to 11 years): Pain, Incapacitating, unable to perform usual activities; Erythema, Swelling, Induration, and Ecchymosis, ≥ 50 mm. Injection site Grade 3 (12 to 17 years): Pain, Significant; prevents daily activity; Erythema, Swelling, Induration, and Ecchymosis, > 100 mm. Systemic Grade 3 (9 to 17 years): Fever, ≥ 39.0°C; Headache, Malaise, Myalgia, and Shivering, Significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site and systemic reactions were analyzed in the Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 100
Percentage of participants
  Injection-site Pain | 56.0
  Grade 3 Injection-site Pain | 0
  Injection-site Erythema | 6.0
  Grade 3 Injection-site Erythema | 0
  Injection-site Swelling | 4.0
  Grade 3 Injection-site Swelling | 0
  Injection-site Induration | 2.0
  Grade 3 Injection-site Induration | 0
  Injection-site Ecchymosis | 1.0
  Grade 3 Injection-site Ecchymosis | 0
  Fever | 0
  Grade 3 Fever | 0
  Headache | 8.0
  Grade 3 Headache | 0
  Malaise | 15.0
  Grade 3 Malaise | 1.0
  Myalgia | 45.0
  Grade 3 Myalgia | 1.0
  Shivering | 3.0
  Grade 3 Shivering | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post vaccination) up to Day 7 post vaccination.
Arm/Group | Quadrivalent Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 56/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent Influenza Vaccine (N=100)
Injection site Pain (General disorders) | 56 (56)
Injection site Erythema (General disorders) | 6 (6)
Headache (Nervous system disorders) | 8 (8)
Malaise (General disorders) | 15 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 45 (45)
Nasopharyngitis (Infections and infestations) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications